CLINICAL TRIAL: NCT00333229
Title: Influence of Zoledronic Acid on Bone Mineral Density and Bone Ultrasonometry in Premenopausal Women With Hormone Receptor Negative Breast Cancer and Adjuvant Chemotherapeutic Treatment
Brief Title: A Study of Zoledronic Acid in the Prevention of Cancer Therapy-induced Bone Loss
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to rare patient population, planned number of patients could not be recruited in a reasonable timeframe. Recruitment was stopped prematurely.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446GDE13; 2004-002831-14
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Primary Hormone Receptor Negative Breast Cancer in Premenopausal Women
Keywords: Breast Cancer; premenopausal; Bone Mineral density; Cancer therapy induced bone loss; zoledronic acid
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic Acid (Experimental): Patients randomized into the Zometa arm received a total of 8 study drug infusions which were applied every 3 months. Patients received treatment for 24 months every 3 months.
  Interventions: Drug: Zoledronic Acid
- Placebo (Placebo Comparator): Patients randomized into the Placebo Arm received a total of 8 placebo infusions which were applied every 3 months. Patients received treatment for 24 months every 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid — 4 mg zoledronic acid in 5 mL concentrate solution. Plastic vials.
  Arms: Zoledronic Acid
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
Breast cancer and osteoporosis are two of the most frequent diseases in women. Estrogen may be associated with bone loss and the risk of breast cancer because of its potent effects on the mitotic activity of breast epithelium and on bone turnover.

This study is will assess the safety and efficacy of Zoledronic acid 4 mg, given every 3 months over 24 months, in improving bone mineral density in premenopausal women with hormone receptor negative breast cancer and adjuvant chemotherapeutic treatment compared to placebo.

This study is not recruiting patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically confirmed incident invasive breast cancer (T1-4) with no evidence of regional lymph node metastasis (N0) or distant metastasis (M0) and after complete primary tumor resection and axillary lymph node dissection less than 90 days before start of study drug treatment.
* Hormone receptor status is negative
* Patient is premenopausal (spontaneous and regular menses with premenopausal estradiol levels (>10ng/dL)
* Patient receives adjuvant standard chemotherapy with approved cytotoxic chemotherapeutic drugs (e.g. AC 4-6 cycles) (prior neoadjuvant CT is allowed)
* Bone density at study entry > -2.5 T-Score

Exclusion Criteria:

* Prior treatment with bisphosphonates and estrogens or treatments for osteoporosis in addition to calcium and vitamin D
* Severe physical or psychological concomitant diseases and other known concurrent, severe medical disorder jeopardizing the life of the patient in the immediate future (e.g., myocardial infarction in previous six months, angina pectoris despite treatment, uncontrolled severe arterial hypertension, progressive cardiac or respiratory failure)
* Known hypersensitivity to bisphosphonates
* Abnormal renal function
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures and recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Marburg, Germany

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (6.2) | 43.2 (2.6) | 42.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) Measured by DXA at Lumbar Spine (L2-L4) Between Baseline and 24 Months.
Time Frame: 24 months
Population: Analysis was not completed as study was not adequately powered due to premature study termination.
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Bone Mineral Density (BMD) Measured by QUS at os Calcis and Phalanges After 24 Months
Time Frame: 2 years
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Course of Biochemical Markers of Bone Turn Over (FSH, Estradiol (E2), Osteocalcin, PINP, Procollagene-I-peptid, Deoxypyridinoline in Serum)
Time Frame: 2 years
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pathologic Fractures During 24 Month
Time Frame: 2 years
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Development of Metastases as Assessed by X-ray, CT, or MRI During 24 Months and During 60 Months
Time Frame: 2 years
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Zoledronic Acid (N=6)
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Zoledronic Acid (N=6)
TINNITUS (Ear and labyrinth disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 | 0
DRY EYE (Eye disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 2
ASTHENIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1
MUCOSAL DRYNESS (General disorders) | 1 | 0
PAIN (General disorders) | 1 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0
FOLLICULITIS (Infections and infestations) | 1 | 0
FURUNCLE (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 0 | 1
ORAL HERPES (Infections and infestations) | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 2 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOSCLEROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
RHEUMATIC FEVER (Musculoskeletal and connective tissue disorders) | 1 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
AMNESIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
PARAESTHESIA (Nervous system disorders) | 3 | 2
SYNCOPE (Nervous system disorders) | 0 | 1
CONVERSION DISORDER (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 2 | 0
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 1 | 1
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 0 | 1
HOT FLUSH (Vascular disorders) | 2 | 2
LYMPHOEDEMA (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.